CLINICAL TRIAL: NCT03205683
Title: Intraneural Facilitation as a Treatment for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Bryan Tsao, Neurology Chairman, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5170247
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraneural facilitation therapy (Experimental): The intraneural facilitation intervention is a novel manual physical therapy approach with anecdotal evidence in neuropathic pain symptoms through biasing blood flow from an artery through the nutrient vessels into the epineurium of an accompanying nerve. The main concept of intraneural facilitation is the use of two manual holds. The first hold is called facilitation hold and includes putting the contralateral joint in a maximal loose-pack position that is comfortable to the patient. The hypothesis with this initial hold is the nerve will have greater excursion the accompanying artery and the nutrient vessels that are clustered at the joint will be stretched. This stretch may enlarge the opening at the junction of the artery and bridging nutrient vessel, therefore consistently creating a vascular bias into the neural epineurial capillaries. Theoretically, this creates increased epifascicular vascular pressure which may be absent due to epineurial ischemia.
  Interventions: Other: Intraneural facilitation (INF)
- Sham therapy (Sham Comparator): Will be performed by a different therapist than actual INF. The patient will be asked to do the following combination of passive range of motion (PROM) and active ROM activities to promote blood flow in the affected arm Each visit will last about 45 minutes, twice a week for 6 weeks (total 12 sessions).
  Missing > 4 sessions will invalidate subject outcomes.
  Interventions: Other: Sham INF

INTERVENTIONS:
Other: Intraneural facilitation (INF) — INF is a novel non-invasive therapy based on the principle of restoring vascular function at the capillary level in peripheral nerve.
  Arms: Intraneural facilitation therapy
Other: Sham INF — Will be performed by a different therapist than actual INF. The patient will be asked to do the following combination of passive range of motion (PROM) and active ROM activities to promote blood flow in the affected arm.
  Arms: Sham therapy

SUMMARY:
We hypothesize that a standard course of INF can result in significant improvement in CTS as measured by clinical, electrodiagnostic, or ultrasound measures.

DETAILED DESCRIPTION:
INF is a novel non-invasive therapy based on the principle of restoring vascular function at the capillary level in peripheral nerve. his therapy has been shown to improve clinical function in patients with diabetic-associated polyneuropathy, a model for various forms of ischemic neuropathy. CTS is a common condition where regional compression at the wrist results in ischemic focal demyelination of the distal median nerve. This results in sensory dysfunction, pain, and eventually axon loss and weakness if the compression is sufficiently severe and prolonged. Standard therapy for CTS includes wrist splints, regional lidocaine injections, ergonomic adjustments, various forms of occupation therapy, and ultimately surgical release of the carpal tunnel ligament. However, all of these are either temporary in their effect or invasive. The diagnosis of CTS relies on clinical, electrodiagnostic or NCS, and ultrasound methods.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred to the LLUH Neurology Electrodiagnostic Laboratory with electrodiagnostic and clinical evidence of CTS (uni- or bilateral)
2. Ages >18 and < 75 (irrespective of gender)
3. Current use of splints as long as the frequency of treatment is unaltered and onset of use is > 1 week in duration

Exclusion Criteria:

1. Prior carpal tunnel release > 2 years ago
2. The presence of any condition that would prevent NCS from accurately diagnosing CTS (e.g., hereditary polyneuropathy or acquired demyelinating polyneuropathy)
3. Workman's Compensation cases
4. Pregnancy
5. Undergoing conservative or surgical/injection therapy (physical or occupational therapy, injections)
6. Clinically silent CTS in face of positive electrodiagnostic results
7. Sufficiently severe clinical symptoms that warrant more aggressive therapy i.e., carpal injections or release
8. Any confounding medical condition that the investigator deems may adversely affect subject participation or outcomes

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
The Boston CTS Questionnaire symptom severity scale and functional assessment. | change between baseline and one week after completion of INF therapy
  composite measurement of carpal tunnel symptomology (pain and numbness) and functional assessment
The Boston CTS Questionnaire symptom severity scale and functional assessment. | change between week 1 and 3 months after completion of INF therapy
  composite measurement of carpal tunnel symptomology (pain and numbness) and functional assessment

SECONDARY OUTCOMES:
Visual analog scale (VAS) | change between baseline and one week after completion of INF therapy
  an ordinal standardized scale grading pain from 0 (absent) to 10 (greatest)
Visual analog scale (VAS) | change between week 1 and 3 months after completion of INF therapy
  an ordinal standardized scale grading pain from 0 (absent) to 10 (greatest)
Ultrasound | change between baseline and one week after completion of INF therapy
  Reduction in diameter of the median nerve at the wrist or in the distal forearm ratio

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Tsao, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No